CLINICAL TRIAL: NCT01594853
Title: Exercise Study of Function and Pathology for Women With X-ALD
Brief Title: Exercise Study of Function and Pathology for Women With X-linked Adrenoleukodystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: European Leukodystrophy Association (Other)
Responsible Party: Principal Investigator, Kathleen Zackowski, Principal Investigator, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00045673
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Results first posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2017-12

CONDITIONS: X-linked Adrenoleukodystrophy
Keywords: exercise; women; training; rehabilitation; leukodystrophy
MeSH Terms: conditions — Adrenoleukodystrophy; Motor Activity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- exercise (Experimental): Female carriers as well as healthy age and gender matched individuals will participate in an exercise paradigm.
  Interventions: Behavioral: exercise training

INTERVENTIONS:
Behavioral: exercise training — The exercise program uses a local Curves® gym to provide an individualized program of strength and cardiovascular training. The program is expected to be performed for 45 minutes 4-6 days per week.
  Other Names: strengthening; Curves

SUMMARY:
The purpose is to see how X-linked adrenoleukodystrophy (X-ALD) is associated with strength and sensation using MRI, in women with X-ALD. The investigators will also see whether exercise can improve these symptoms for women with X-ALD.

DETAILED DESCRIPTION:
X-linked adrenoleukodystrophy (X-ALD), a [sex-linked] progressive neurodegenerative disease, is caused by a defect in the ABCD1 gene. The disease is expressed in multiple ways, but the most common adult form is adrenomyeloneuropathy (AMN), which results in slowly progressive changes in muscle tone and weakness, sensory loss, and dysfunction of the autonomic nervous system. In a previous study the investigators linked abnormalities in the [brain/spinal cord] to lower extremity weakness in men with AMN; however, there have been no studies evaluating these relationships in women carriers (i.e., women with AMN). It is unknown, in women with AMN, how the pattern of damage in the brain and spinal cord relates to disability and if these patterns predict responsiveness to treatment. The investigators hypothesize that by using magnetization transfer (MT) and diffusion tensor imaging (DTI), two magnetic resonance imaging (MRI) modalities, to track particular changes in the brain and spinal cord will predict disability and additionally, who is likely to respond best to a training regimen. The investigators expect that these more advanced imaging techniques will be more sensitive and accurate quantitative measures of clinical motor function and women with greater loss in the spinal cord compared to the brain will benefit most from training to improve disability. To test this hypothesis, women with AMN will receive MRI scans at baseline and complete measures of global walking and lower extremity impairments of vibration sensation, spasticity, and strength at three time-points: baseline, 12 weeks, and 18 weeks after baseline. The group will participate in a resistive training program for 12 weeks. MRI data will be correlated to changes over time in measures of impairment to determine their relationships. The linking of this information will not only be important for better defining disability in women with AMN but it will also help to guide physicians and rehabilitation therapists in predicting who is likely to respond to rehabilitative interventions, as well as for optimizing the effects of future pharmacological interventions.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis, X-ALD heterozygote carrier
* no medical contraindication to participating in a strength training program
* able to follow complex directions as determined by a score of ≤1 on a subset of questions taken from the NIH Stroke scale (Brott et al. 1989)
* hip flexion strength: 6.6-15.8kg
* hip extension strength: up to 18.3 kg
* normal passive range of motion at hips/knees/ankles
* able to walk ≥50m

Exclusion Criteria:

* Evidence of other neurological deficit that could interfere, such as previous stroke or muscle disease
* congestive heart failure
* cancer
* orthopedic conditions
* severe pain that precludes study participation
* seizures
* pregnancy
* other medical condition that precludes participation in an exercise program, e.g., unstable angina, uncontrolled diabetes, uncontrolled hypertension

Healthy controls have the same age and exclusion criteria as women with AMN except that they will not be carriers for X-ALD. They must have normal neurological function.

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Zackowski, Ph.D., Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Motion Analysis Lab, Baltimore, Maryland, United States

REFERENCES:
- See also: See Clinical Research Projects listing. — http://www.kennedykrieger.org/research-training

RESULTS

PARTICIPANT FLOW:
Groups:
- Female Carriers: Female carriers will participate in an exercise paradigm.
  exercise training: The exercise program uses a local Curves® gym to provide an individualized program of strength and cardiovascular training. The program is expected to be performed for 45 minutes 4-6 days per week.
- Healthy Controls: Healthy age and gender matched individuals will participate in an exercise paradigm.
  exercise training: The exercise program uses a local Curves® gym to provide an individualized program of strength and cardiovascular training. The program is expected to be performed for 45 minutes 4-6 days per week.
Period: Overall Study
Arm/Group | Female Carriers | Healthy Controls
Started | 16 | 15
Completed | 14 | 12
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — noncompliance with exercise | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Female Carriers | Healthy Controls | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (8.4) | 51.3 (12.5) | 51.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 13 | 9 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximal Voluntary Contraction of the Hip Flexors From Baseline to End of Training and to Post-training
Description: Here, we will assess whether the degree of a person's white matter integrity (i.e. for tracts of interest as measured from MRI) predicts their ability to benefit from exercise. Our prediction is that those individuals with preserved white matter integrity will show the greatest improvement in hip flexor strength.
Time Frame: Participants are assessed at baseline (visit 1, enrollment), end of training (visit 2, week 12) and post-training (visit 3, week 18).
Population: For the follow up visit, there are fewer participants in the analysis because 5 female carriers and 1 control were unable to return for the third follow up visit due to burden to travel costs.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Female Carriers | Healthy Controls
Number analyzed (Participants) | 14 | 12
kg
  Change post-training | 0.94 (1.14) | 0.98 (2.01)
  Change at follow up: number analyzed (Participants) | 11 | 9
  Change at follow up | 1.32 (1.28) | 1.37 (1.68)

ADVERSE EVENTS:
Arm/Group | Female Carriers | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 0/14 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-07-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT01594853/Prot_SAP_000.pdf